CLINICAL TRIAL: NCT00168662
Title: Trial of Two-Dose Standard Measles Vaccination Schedule: Long-Term Impact on Morbidity and Mortality of a Two-Dose Vaccination Schedule at 6 and 9 Months of Age Compared With a Standard Regimen of One Dose at 9 Months of Age
Brief Title: Non-Specific Effects of Standard Titre Measles Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: International Cooperation with Developing Countries (Other); Danish Council for Development Research (Other); Medical Research Council Unit, The Gambia (Other)
Responsible Party: May-Lill Garly, Bandim Health Project
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC18-CT95-0011-Twodose1; EU grant: IC18-CT95-0011
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-02

CONDITIONS: Measles
Keywords: Non-specific effects of vaccines; Infant mortality; Child mortality; Mortality; Morbidity; Measles vaccine; Measles; Immunisation; Low income country; Guinea-Bissau; Bandim Health Project; Immunology
MeSH Terms: conditions — Measles; Infant Death | interventions — Poliovirus Vaccine, Inactivated

INTERVENTIONS:
Biological: Measles and inactivated polio vaccine

SUMMARY:
The general objectives of the proposed research work are:

A1) to reduce childhood mortality in developing countries through better control of measles infection by finding the best immunization strategy, and A2) to investigate the hypothesis that standard titre measles immunization is associated with non targeted beneficial effects on childhood morbidity and mortality in developing countries.

The measurable, specific objectives of the present proposal are:

B1) to examine whether a two-dose strategy for measles immunization at 6 and 9 months of age can reduce measles incidence by 50% through better coverage or improved seroconversion, and B2) to examine whether a two-dose strategy for measles immunization at 6 and 9 months of age can reduce childhood mortality by 20% through better coverage, better protection against measles or non targeted beneficial effects, and B3) to determine the magnitude and duration of non-measles related changes in morbidity patterns after standard titre measles immunization, in particular to test whether measles immunization is associated with a 15% reduction in the risk of diarrhoea, and B4) to determine non-measles related immunological changes among recipients of measles vaccine in order to establish possible pathways for the non targeted effects of standard titre measles immunization.

DETAILED DESCRIPTION:
Background. Measles is the major killer among vaccine preventable diseases with an estimated one million deaths/year in developing countries. Though a good vaccine exists, the current immunization strategy of one dose at 9 months is far from optimal; too many children get measles before the age of immunization, coverage is too low when immunization has to wait until 9 months of age, and the protective efficacy is insufficient with the current vaccine given at 9 months of age. There is therefore a need for alternative immunization strategies or new vaccines.

Evaluations of vaccines have usually been based on a disease specific perspective; i.e. evaluation of specific immunity, and protective efficacy against the specific disease, its complications and mortality. However, our research from Guinea-Bissau, Senegal and Bangladesh has indicated that measles immunization and measles infection may have non-specific beneficial effects. The present protocol is an attempt to assess the magnitude and possible mechanisms of the non targeted beneficial effects of measles immunization and measles infection as well as an attempt to assess some of the practical implications of the hypothesis about non-specific beneficial effects.

Approach and methodologies. We tested a two dose measles immunization strategy at 6 and 9 months compared with the currently recommended strategy of one dose at 9 months. The children were be randomized to receive measles immunization at 6 and 9 months of age or inactivated polio at 6 months and measles at 9 months of age.

The non targeted effects of measles immunization on mortality and morbidity are best studied within a randomized trial comparing immunized and unimmunized children. In order to study the impact on non-measles related morbidity, some children recruited for the immunization trial will be included in weekly morbidity surveillance for diarrhoea, respiratory infections and malaria which are the most important disease complexes for childhood mortality in Guinea-Bissau.

Possible immunological differences between measles immunized and unimmunized children will be examined through measurements of T-lymphocyte levels, neopterin, beta2-microglobulin, delayed hypersensitivity (Multitest), allergic reactions (skin prick tests), antibody responses to other antigens (tetanus) and thymus growth (by sonography). Functional differences will be tested by response to a second vaccine antigen (HBV) at 7½ and 9 months of age when only one group has received measles vaccine.

ELIGIBILITY:
Inclusion Criteria: Infants of 6 months of age registered in the Bandim Health Project registration system and currently living in the Bandim Health Project areas: Bandim I, Bandim II, Belem and Mindará

Exclusion Criteria: Severe illness requiring hospitalisation

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7800
Dates: Start 1995-03; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Vaccination coverage
Vaccine efficacy
Measles specific mortality
All cause mortality until 3 years of age

SECONDARY OUTCOMES:
Measles antibodies at 6, 7½, 9, 10½ and 18 months of age
T-cells at 6, 7½, 9, 10½ and 18 months of age
Thymus size at 6, 7½, 9, 10½ months of age
Neopterin level at 7½ months of age
Beta-2-microglobulin level at 7½ months of age
Hepatitis B antibodies at 7½, 9 and 10½ months of age
Tetanus antibodies at 9 months og age
Delayed type hypersensitivity at 7½ months of age
Skin prick test (allergy) at 7½ months of age
Morbidity from 6 to 18 months of age
Anthropometric measures at 6, 7½, 9, 10½ and 18 months of age

CONTACTS AND LOCATIONS:
Overall Officials: PETER AABY, MSc, Dr. Med, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Apartado 861, Guinea-Bissau

REFERENCES:
- [Background] Veirum JE, Sodemann M, Biai S, Jakobsen M, Garly ML, Hedegaard K, Jensen H, Aaby P. Routine vaccinations associated with divergent effects on female and male mortality at the paediatric ward in Bissau, Guinea-Bissau. Vaccine. 2005 Jan 19;23(9):1197-204. doi: 10.1016/j.vaccine.2004.02.053. PMID 15629363
- [Result] Garly ML, Martins CL, Bale C, da Costa F, Dias F, Whittle H, Aaby P. Early two-dose measles vaccination schedule in Guinea-Bissau: good protection and coverage in infancy. Int J Epidemiol. 1999 Apr;28(2):347-52. doi: 10.1093/ije/28.2.347. PMID 10342702
- [Result] Garly ML, Bale C, Martins CL, Monteiro M, George E, Kidd M, Dias F, Aaby P, Whittle HC. Measles antibody responses after early two dose trials in Guinea-Bissau with Edmonston-Zagreb and Schwarz standard-titre measles vaccine: better antibody increase from booster dose of the Edmonston-Zagreb vaccine. Vaccine. 2001 Feb 28;19(15-16):1951-9. doi: 10.1016/s0264-410x(00)00431-x. PMID 11228365
- [Result] Garly ML, Bale C, Martins CL, Balde MA, Hedegaard KL, Whittle HC, Aaby P. BCG vaccination among West African infants is associated with less anergy to tuberculin and diphtheria-tetanus antigens. Vaccine. 2001 Nov 12;20(3-4):468-74. doi: 10.1016/s0264-410x(01)00339-5. PMID 11672911
- [Result] Aaby P, Jensen H, Garly ML, Bale C, Martins C, Lisse I. Routine vaccinations and child survival in a war situation with high mortality: effect of gender. Vaccine. 2002 Nov 22;21(1-2):15-20. doi: 10.1016/s0264-410x(02)00441-3. PMID 12443658
- [Result] Garly ML, Martins CL, Bale C, Balde MA, Hedegaard KL, Gustafson P, Lisse IM, Whittle HC, Aaby P. BCG scar and positive tuberculin reaction associated with reduced child mortality in West Africa. A non-specific beneficial effect of BCG? Vaccine. 2003 Jun 20;21(21-22):2782-90. doi: 10.1016/s0264-410x(03)00181-6. PMID 12798618
- [Result] Aaby P, Garly ML, Bale C, Martins C, Jensen H, Lisse I, Whittle H. Survival of previously measles-vaccinated and measles-unvaccinated children in an emergency situation: an unplanned study. Pediatr Infect Dis J. 2003 Sep;22(9):798-805. doi: 10.1097/01.inf.0000083821.33187.b5. PMID 14506371
- [Result] Aaby P, Jensen H, Rodrigues A, Garly ML, Benn CS, Lisse IM, Simondon F. Divergent female-male mortality ratios associated with different routine vaccinations among female-male twin pairs. Int J Epidemiol. 2004 Apr;33(2):367-73. doi: 10.1093/ije/dyh004. PMID 15082642
- [Result] Garly ML, Jensen H, Martins CL, Bale C, Balde MA, Lisse IM, Aaby P. Hepatitis B vaccination associated with higher female than male mortality in Guinea-bissau: an observational study. Pediatr Infect Dis J. 2004 Dec;23(12):1086-92. PMID 15626943
- [Result] Roth A, Gustafson P, Nhaga A, Djana Q, Poulsen A, Garly ML, Jensen H, Sodemann M, Rodriques A, Aaby P. BCG vaccination scar associated with better childhood survival in Guinea-Bissau. Int J Epidemiol. 2005 Jun;34(3):540-7. doi: 10.1093/ije/dyh392. Epub 2005 Jan 19. PMID 15659474
- See also: Statens Serum Institut, Denmark — http://www.ssi.dk